CLINICAL TRIAL: NCT04885660
Title: Bioequivalence Study of Compound Lisinopril Tablets
Brief Title: Bioequivalence Evaluation of Two Fixed-dose Combination of Lisinopril 10mg/Levamlodipine Besylate 5mg in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SR-BE-001
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Therapeutic Equivalency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compound lisinopril tablets (Experimental): a single oral of Compound lisinopril tablets test formulation( Lisinopril 10mg/Levamlodipine besylate 5mg)
  Interventions: Drug: compound lisinopril tablet
- Compound lisinopril tablets(Lisonorm®) (Active Comparator): a single oral of Compound lisinopril tablets reference formulation( Lisinopril 10mg/Levamlodipine besylate 5mg)
  Interventions: Drug: compound lisinopril tablet(Lisonorm®)

INTERVENTIONS:
Drug: compound lisinopril tablet — The subjects randomly received single oral administration of compound lisinopril tablet(Lisinopril 10mg/Levamlodipine besylate 5mg)
  Arms: Compound lisinopril tablets
Drug: compound lisinopril tablet(Lisonorm®) — The subjects randomly received single oral administration of compound lisinopril tablet(Lisonorm®)
  Arms: Compound lisinopril tablets(Lisonorm®)

SUMMARY:
The bioavailability of compound lisinopril tablets (specification: lisinopril 10mg / amlodipine 5mg) developed by Sichuan shangrui biomedical Co., Ltd. was compared with that of reference compound lisinopril tablets (specification: lisinopril 10mg / amlodipine 5mg) produced by Hungary Gedeon Richter Pharmaceutical Co., Ltd.The bioequivalence of single dose of test preparation and reference preparation was evaluated in heathy subjects under fasting and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

- 1.Healthy male and female aged over 18years 2.Subjects willing to provide written informed consent and to adhere to protocol requirements 3.Subject's weight within normal range according to normal values for Body Mass Index (19.00 to 26.00 kg/m2 (both inclusive)), males with minimum of 50 kg weight, females with minimum of 45kg weight.

4.Subjects have not clinically significant abnormalities, including vital signs, physical examinations, laboratory tests, and ECG as determined by clinical examination

Exclusion Criteria:

* 1.History or presence of significant cardiovascular, Urogenital, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder 2.Allergic constitution(Allergic to two or more substances) or hypersensitivity to investigational product 3.History or presence of significant gastrointestinal inflammation /ulcer. or other medical history affecting drug absorption 4.Use of any drugs or herbal medicine within 14 days prior to the first dose 5.Can not follow approved birth control methods (a double barrier method) from the screening（Female subjects from two weeks prior to the screening） till 3 months after the last dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 90 days
  Evaluate the Cmax of Lenopril and amlodipine for test preparation and reference preparation

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li T, Liu YP, Liu SQ, Shi P, Jiang X, Tao Y, Gao XM, Ma YP, Cao Y. Bioequivalence evaluation and food effect assessment of Lisinopril/amlodipine tablets in healthy Chinese subjects under fasting and fed conditions. BMC Pharmacol Toxicol. 2022 Jul 7;23(1):45. doi: 10.1186/s40360-022-00590-6. PMID 35794660